CLINICAL TRIAL: NCT03743259
Title: A Multicenter, Open-label, Parallel, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of LuminoMark Inj. (Conc. for Fluorescence) Localization in Patients With Nonpalpable Breast Lesions
Brief Title: To Evaluate the Efficacy and Safety of LuminoMark Injection in Patients With Nonpalpable Breast Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL_LMN_201
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-01

CONDITIONS: Breast Diseases
Keywords: Nonpalpable Breast Lesions
MeSH Terms: conditions — Breast Diseases | interventions — Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LuminoMark inj. 0.1mL (Experimental): Injection LuminoMark inj. 0.1mL once in this study.
  Interventions: Drug: LuminoMark inj. 0.1mL
- LuminoMark inj. 0.2mL (Experimental): Injection LuminoMark inj. 0.2mL once in this study.
  Interventions: Drug: LuminoMark inj. 0.2mL
- Charcotrace Inj. (Active Comparator): Charcotrace Inj. about 0.3~1mL
  Interventions: Drug: Charcotrace Inj.

INTERVENTIONS:
Drug: LuminoMark inj. 0.1mL — Injection LuminoMark inj. (Conc. for fluorescence) 0.1mL once in this study.
  Other Names: LuminoMark inj.(Conc. for fluorescence) 0.1mL
  Arms: LuminoMark inj. 0.1mL
Drug: LuminoMark inj. 0.2mL — Injection LuminoMark inj. (Conc. for fluorescence) 0.2mL once in this study.
  Other Names: LuminoMark inj.(Conc. for fluorescence) 0.2mL
  Arms: LuminoMark inj. 0.2mL
Drug: Charcotrace Inj. — Injection Charcotrace Inj. about 0.3~1mL once in this study.
  Other Names: Charcotrace Injection(Activated Charcoal 40mg/1ml)
  Arms: Charcotrace Inj.

SUMMARY:
This study is a multicenter, Open-label, Parallel, Phase 2 Clinical Trial in 6 weeks for screening, once Investigational product injection, Follow up visit.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of LuminoMark inj. (Conc. for fluorescence) localization in patients with nonpalpable breast lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 19 years ≤ age ≥ 80 years
2. Those who be expected to do operation about non palpable breast lesion excision
3. Those who have lesion vial mammography and breast ultrasound
4. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients who be expected to do mastectomy
2. Patients with multiple tumor or diffuse microcalcification
3. Patients who have ink on invasive cancer or ductal carcinoma in situ despite 3 times local resection
4. Patients who were treated with moderate to severe radiotherapy
5. Patients who were treated with neoadjuvant Chemotherapy
6. Patients with active invading skin connective tissue disease
7. Patients with local progressing breast cancer or inflammatory local progressing breast cancer
8. Patients who have an allergy to investigational product or any of the component with the Investigational product
9. Patients who disagree about contraception for this clinical trial
10. A pregnant women or lactating women
11. Patients who participated in other clinical trials within the past 12 weeks from the date of informed consent
12. Patients who investigators determines unsuitable for this clinical trial

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female
Enrollment: 44 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Excision perfection(It is a formula. This formula's calculation method is as follows. [Excision perfection = the longest diameter of removed lesion after surgery / the longest diameter of identified lesion via breast ultrasonography results]) | Visit 3(Day 0)
  Excision perfection is how well the surgeon removed the lesion compared to an identified by breast ultrasonography. Visit 3, Investigators calculate 'Excision perfection' using by the formula.

SECONDARY OUTCOMES:
Coloring confirmation rate of excision lesion. | Visit 3(Day 0)
  The proportion of colored excision lesion
Technical success rate | Visit 3(Day 0)
  The proportion of colored lesion when make an incision
Pathologic perfection(It is a formula. This formula's calculation method is as follows. [Pathologic perfection = the longest diameter of measured lesion by gross(=visual) pathologic method / the longest diameter of removed lesion after surgery]) | Visit 3(Day 0)
  Pathologic perfection is how well the surgeon removed the lesion compared to an identified by gross pathologic method. Visit 3, Investigators calculate 'Pathologic perfection' using by the formula.
Pigmentation | Visit 5(Day 10~Day 24)
  Check whether skin is pigmented or not

CONTACTS AND LOCATIONS:
Overall Officials: Seok Won Kim, PI, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim I, Choi HJ, Ryu JM, Lee SK, Yu JH, Lee JE, Nam SJ, Shin HJ, Kim SW. The efficacy and safety of indocyanine green-hyaluronic acid mixture (LuminoMark) for localization in patients with non-palpable breast lesions: a multi-center open-label parallel phase-2 clinical trial. BMC Surg. 2021 Mar 16;21(1):134. doi: 10.1186/s12893-021-01129-y. PMID 33726718